CLINICAL TRIAL: NCT05707663
Title: Longitudinal Assessment of Brain Structure and Function in Juvenile Onset Huntington's Disease (JoHD)
Brief Title: Longitudinal Assessment of Brain Structure and Function in Juvenile-onset Huntington's Disease
Status: Recruiting | Type: Observational
Sponsor: University of Iowa (Other)
Collaborators: Columbia University (Other); University of California, Davis (Other); The University of Texas Health Science Center, Houston (Other); Children's Hospital of Philadelphia (Other); George-Huntington-Institut GmbH (Other); UCL Queen Square Institute of Neurology (Other)
Responsible Party: Principal Investigator, Peggy C Nopoulos, Professor, University of Iowa
Other Study IDs: 201109879
Record Dates: First submitted 2022-12-16; First posted 2023-02-01 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2024-12

CONDITIONS: Juvenile Huntington Disease; Juvenile-Onset Huntington Disease
Keywords: JoHD; JHD; Juvenile Huntington Disease; Juvenile Huntington's Disease; Juvenile-onset Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Bio-specimens are collected and retained for all participants for future research. Specimens are a single sample of 3-4 teaspoons of blood drawn from the arm that consist of whole blood, plasma and DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- JoHD: Children adolescents and young adults ages 6-30 who have been clinically diagnosed with Juvenile-onset Huntington's Disease

SUMMARY:
The goal of this observational study is to learn about brain development in Juvenile-onset Huntington's Disease (JoHD). The main questions it aims to answer are:

* Is brain development different in JoHD than Adult-onset Huntington's Disease (AoHD)?
* Can reliable biomarkers for JoHD be found in brain structure and function?

Participants will be asked to complete cognitive tests, behavioral assessments, physical and neurologic evaluation, and MRI. Data collected will be compared to populations who are at-risk for HD and who have been diagnosed with HD as adults.

DETAILED DESCRIPTION:
Huntington's disease (HD) is a genetic neurodegenerative disorder caused by an abnormal expansion of a trinucleotide CAG repeat region of the huntingtin gene (HTT). The majority of patients with HD do not present with symptoms until the age of 40-50 years old, on average, which is referred to as Adult-onset HD (AoHD). A much smaller percentage of patients with HD receive a motor diagnosis prior to the age of 21, which is referred to as Juvenile-onset HD (JoHD). Although patients with JoHD have the same core triad of cognitive, behavior, and motor symptoms, there are unique clinical characteristics that are distinct from AoHD. Specifically, patients with JoHD have less chorea compared to patients with AoHD, often presenting with rigidity and bradykinesia. However, due to the rarity, there is a lack of data regarding symptom characterization, neurobiology and progression of JoHD. Large-scale observational studies have been performed in AoHD, which have broadened our understanding of HD and opened the doors for the development and conduct of clinical trials. Patients with JoHD have been excluded from clinical trials, leaving patients and their families feeling hopeless and abandoned by the scientific community. Large-scale, longitudinal studies in patients with JoHD are critical to bettering our understanding of this devastating disease and providing hope to patients who have felt left behind as therapeutic strategies advance in AoHD.

In an effort to better understand the developmental aspects of this brain disease, the current study proposes to evaluate brain structure and function in children, adolescents, and young adults (ages 6-30) who have been diagnosed with JoHD. Brain structure will be evaluating using Magnetic Resonance Imaging (MRI) with quantitative measures of the entire brain, cerebral cortex, as well as white matter integrity via Diffusion Tensor Imaging. Brain function will be assessed by cognitive tests, behavioral assessment, and physical and neurologic evaluation. This study will test the hypothesis that comprehensive and longitudinal assessments of brain function and brain structure may produce reliable biomarkers of disease progression in JoHD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of JoHD
* Aged 6-30

Exclusion Criteria:

* Metal in body
* History of head trauma, brain tumor, seizures or epilepsy unrelated to JoHD
* History of major surgery or serious chronic medical conditions other than JoHD

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, adolescents and young adults ages 6-30 who have been clinically diagnosed with Juvenile-onset Huntington's Disease
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Volume of brain structures as measured by Magnetic Resonance Imaging (MRI) | 60-90 minutes out of 7-8 hour testing day
  Magnetic Resonance Imaging (MRI) and Diffusion Tensor Imaging (DTI) data will be analyzed to assess brain structure based upon variables including global volume, total cerebral spinal fluid, subregion volumes, cortical surface anatomy including cortical depth, surface area and gyral shape, and symmetry between brain hemispheres.

SECONDARY OUTCOMES:
Quantitative assessment of cognitive skills and behavioral factors | 5 hours out of 7-8 hour testing day
  Participants undergo a cognitive battery which will quantify skills such as attention, learning, memory. In addition, behavioral measures will be administered in both self and proxy report formats.

OTHER OUTCOMES:
Quantitative assessment of motor performance | 1 hour out of 7-8 hour testing day
  Motor skill (both fine and gross) will be assessed and quantified via standard UHDRS motor exam and Q-Motor/Q-Cog equipment suite.
Quantification of Neurofilament Light | 10 minutes for blood draw out of 7-8 hour testing day
  Plasma samples will be sent for each visit to University College of London for analysis of NfL, an indicator of neuronal damage determine viability as a biomarker for Huntington's Disease.
Demographic and Physiological Data | 10 minutes for vitals collection out of 7-8 hour testing day
  Analyses will control for age, sex and height/weight. Age will be recorded in whole months. Sex will be recorded as gender assigned at birth with current gender identity noted. Height will be measured in centimeters, and weight will be measured in kilograms.

CONTACTS AND LOCATIONS:
Overall Officials: Peggy C Nopoulos, MD, Principal Investigator — University of Iowa
Locations (6):
- United States (6):
  - University of California Davis, Sacramento, California
  - University of Iowa Hospitals and Clinics, Department of Psychiatry, Iowa City, Iowa
  - Columbia University Medical Center, New York, New York
  - Children's Hospital of Philadelphia with the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Aggregate, de-identified data may be shared with approved collaborators, but individual participant data will not be shared.

REFERENCES:
- [Result] Nopoulos PC. Special Issue: Juvenile Onset Huntington's Disease. Brain Sci. 2020 Sep 20;10(9):652. doi: 10.3390/brainsci10090652. PMID 32962249
- See also: Study site — http://kids-johd.org
- See also: Study site — http://www.facebook.com/johdbrainstudy
- See also: Study site — http://mobile.twitter.com/johd_iowa